CLINICAL TRIAL: NCT06089733
Title: a Single-center, Open-label, Fixed Sequence Study in Healthy Chinese Subjects to Evaluate the Pharmacokinetic Effects of Itraconazole and Rifampicin on Oral Administration of a Single Dose of ABSK021
Brief Title: A Clinical Trial to Evaluate the Effect of Itraconazole and Rifampicin on ABSK021
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK021-103
Record Dates: First submitted 2023-06-13; First posted 2023-10-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Intervention Model Description: On Day 1, subjects will receive a single oral dose of approximately 50 mg ABSK021 containing approximately 100 μCi of [14C] ABSK021 in the fasted state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABSK201 and Itraconazole/Rifampicin (Experimental): Part A: Subjects will receive a single 10mg Oral administration of ABSK021 at C1D1, followed by a washout period of at least 14 days. The second cycle (C2): after the end of the first cycle, the subjects will receive 200 mg of C2D1-C2D24 Itraconazole oral liquid and a single 10 mg of ABSK021 Oral administration at C2D4.
  Part B: Subjects will receive a single dose of 50 mg of ABSK021 Oral administration once at C1D1, followed by a washout period of at least 14 days. Subjects will receive 600 mg of Rifampicin capsules once a day at C2D1-C2D15 and a single dose of ABSK021 Oral administration at C2D7, with the dose of 50 mg.
  Interventions: Drug: Part A ABSK201 and Itraconazole; Drug: Part A ABSK201 and Rifampicin

INTERVENTIONS:
Drug: Part A ABSK201 and Itraconazole — Subjects will receive a single 10mg Oral administration of ABSK021 at C1D1, followed by a washout period of at least 14 days. The second cycle (C2): after the end of the first cycle, the subjects will receive 200 mg of C2D1-C2D24 Itraconazole oral liquid and a single 10 mg of ABSK021 Oral administration at C2D4.
Drug: Part A ABSK201 and Rifampicin — Subjects will receive a single dose of 50 mg of ABSK021 Oral administration once at C1D1, followed by a washout period of at least 14 days. Subjects will receive 600 mg of Rifampicin capsules once a day at C2D1-C2D15 and a single dose of ABSK021 Oral administration at C2D7, with the dose of 50 mg.

SUMMARY:
This study is a single center, open lable and fixed sequence test conducted in healthy subjects to evaluate the pharmacokinetic effects of Itraconazole and Rifampicin on a single dose of ABSK021 Oral administration. It is planned to enroll 32 healthy subjects and assign them to two parallel test groups, Part A (ABSK021 combined with Itraconazole) and Part B (ABSK021 combined with Rifampicin).

DETAILED DESCRIPTION:
Each study section includes a screening period conducted within 28 days prior to the first administration of the investigational drug, a trial period of 2 cycles, and withdrawal visits on the 21st or 14th day (Part A) or 14th day (Part B) after the last dose of ABSK021. This study will end after all participants complete 2 cycles of the trial period and withdraw from the study visit.

Whether subjects who have completed the first cycle of the study will enter the second cycle of the study will be determined by the researcher based on their physical condition and relevant visit examination results. For the subjects who interrupted or permanently suspended the study due to adverse events or clinically significant laboratory Outlier, the interview rate shall be determined according to the requirements of the research institution or the clinical indication syndrome until the AE is resolved or stabilized, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 18 and 45 years old (including 18 and 45 years old) during screening, with no less than 6 single gender subjects in each group;
* Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) between 19 and 28 (including 19 and 28), BMI=weight (kg)/height (m) ^2;
* Medical history, physical examination, clinical laboratory examination, and other relevant examinations before screening that have been determined by the researcher to be normal or abnormal without clinical significance;
* Male or female subjects with Fertility must agree to use an effective contraceptive method (see 5.4 for details) during the study period and within 6 months after the last dose of test drug administration, and male subjects will not donate sperm during this period; Female subjects must be non pregnant and non breast-feeding female subjects. Pregnancy is defined as women who are pregnant until the termination of pregnancy. It is determined by the laboratory hCG test within 7 days before the start of the study;
* Voluntarily participate in this clinical trial, understand the research procedure, and sign an informed consent form before screening; Good compliance and willingness to follow research procedures.

Exclusion Criteria:

* If there is a history of cardiovascular, respiratory, blood, liver, kidney, gastrointestinal, endocrine or Nervous system disease diseases, the absorption, metabolism or elimination of drugs are significantly affected, and the investigator judges that the use of experimental drugs may pose risks, interfere with the interpretation of data or affect the ability of subjects to participate in the study;
* Known or persistent mental disorders that may interfere with the participant's participation in the study, as determined by the researcher;
* Known to have a history of allergy to food, experimental drug ABSK021, Rifampicin, Itraconazole or other drugs;
* Those who have participated in drug clinical trials as subjects within the past 3 months;
* I have previously participated in this study or any other studies related to ABSK021 as a subject and have taken ABSK021.
* Those who have applied CYP3A4 strong inhibitor or inducer within 14 days before the first administration (including Grapefruit juice, Grapefruit hybrids, pomegranate, carambola, grapefruit, seville orange, juice or other processed products);
* There are factors that significantly affect the absorption, distribution, metabolism and excretion of drugs, such as inability to take test drugs orally, obvious nausea, vomiting and Malabsorption;
* Those who are unwilling to comply with the dietary requirements/restrictions during the study period, the specific dietary requirements are: (i) only consume the meals provided by the research center during hospitalization, (ii) avoid consuming CYP3A4 strong inhibitors or inducers during the study period;
* Within the first 3 months of screening, those who consume more than 14 units of alcohol per week (1 unit of alcohol is approximately 360mL of beer or 45mL of 40% alcohol or 150mL of wine), or who are positive for alcohol screening, or are unwilling to comply with the alcohol restrictions specified in section 5.3.3;
* Smoking at least 5 cigarettes per day (or corresponding amounts of tobacco or nicotine products) within the first 3 months of screening; Or those who are unwilling to comply with the smoking restrictions specified in Section 5.3.3;
* The researcher judged that there were people who had excessive intake of methyl Xanthine/caffeine in the past 6 months (excessive intake is defined as more than 6 units of caffeine per day, and 1 unit of caffeine is equivalent to 177 milliliters of coffee, 355 milliliters of tea, 355 milliliters of cola, or 85 grams of chocolate), or were unwilling to comply with the restrictions on the use of methyl Xanthine/caffeine in 5.3.3 during the study period;
* People with positive serum hepatitis B B surface antigen (HBsAg), hepatitis B B e antigen (HBeAg), hepatitis B B e antibody (HBeAb), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody, HIV (HIV) antibody screening;
* Those with a history of bacterial, fungal, parasitic, viral (excluding nasopharyngitis, COVID-19), mycobacterial infection, or clinically significant abnormal chest X-ray results within 45 days before the first administration (determined by the investigator);

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Part A_(1)Pharmacokinetic Outcome Measures of ABSK021 after single oral administration of ABSK021 capsules and combination of itraconazole oral solution using Peak Plasma Concentration (Cmax) | Conduct testing within 1 month after all volunteers collect PK samples at all time points required by the protocol
  Collect plasma samples of ABSK021 and its metabolites (if data allows), as well as itraconazole and its metabolite hydroxyitraconazole, from all subjects before and after administration for PK evaluation. Plasma samples of ABSK021 and its metabolites (if data allows) are collected at C1 and C2, while plasma samples of itraconazole and its metabolite hydroxyitraconazole are collected at C2.
Part A_(2)Pharmacokinetic Outcome Measures of ABSK021 after single oral administration of ABSK021 capsules and combination of itraconazole oral solution using Area under the plasma concentration versus time curve (AUC) | Conduct testing within 1 month after all volunteers collect PK samples at all time points required by the protocol
  Collect plasma samples of ABSK021 and its metabolites (if data allows), as well as itraconazole and its metabolite hydroxyitraconazole, from all subjects before and after administration for PK evaluation. Plasma samples of ABSK021 and its metabolites (if data allows) are collected at C1 and C2, while plasma samples of itraconazole and its metabolite hydroxyitraconazole are collected at C2.
Part B_(1)Pharmacokinetic Outcome Measures of ABSK021 after single oral administration and in combination with Rifampicin using Peak Plasma Concentration (Cmax). | Conduct testing within 1 month after all volunteers collect PK samples at all time points required by the protocol
  Collect plasma samples of ABSK021 and its metabolites (if data allows) and rifampicin from all subjects before and after administration for PK evaluation. Plasma samples of ABSK021 and its metabolites (if data allows) are sampled at C1 and C2, while rifampicin plasma samples are sampled at C2.
Part B_(2)Pharmacokinetic Outcome Measures of ABSK021 after single oral administration and in combination with Rifampicin using Area under the plasma concentration versus time curve (AUC). | Conduct testing within 1 month after all volunteers collect PK samples at all time points required by the protocol
  Collect plasma samples of ABSK021 and its metabolites (if data allows) and rifampicin from all subjects before and after administration for PK evaluation. Plasma samples of ABSK021 and its metabolites (if data allows) are sampled at C1 and C2, while rifampicin plasma samples are sampled at C2.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Professor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No